CLINICAL TRIAL: NCT06084988
Title: An Open-Label Single-Arm Phase I/IIa Study to Evaluate the Safety of Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product StromaForte for the Treatment of Knee Osteoarthritis
Brief Title: A Study to Evaluate the Safety of Human Allogeneic Bone-Marrow-Derived Mesenchymal Stromal Cell Product StromaForte for the Treatment of Knee Osteoarthritis
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Cellcolabs Clinical SPV Limited (Industry)
Collaborators: PDC-CRO (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 00-OA Study-2022
Record Dates: First submitted 2023-10-11; First posted 2023-10-16 (Actual); Last update posted 2023-11-22 (Actual); Status verified 2023-11

CONDITIONS: Osteo Arthritis Knee

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MSC Intervention Group (Experimental): Participants will receive one dose (50 x 106 allogeneic bone marrow (BM)-derived MSC formulated in 4 ml infusion solution (sodium chloride supplemented with human serum albumin) to be given via ultrasound-guided intra-articular injection of human allogeneic bone marrow-derived mesenchymal stromal cell product StromaForte. All patients will be observed for at least 2 hours post-injection at the study site. Both active monitoring and spontaneous reporting will be used.
  Interventions: Biological: Human Allogenic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte)

INTERVENTIONS:
Biological: Human Allogenic Bone-Marrow-Derived Mesenchymal Stromal Cell Product (StromaForte) — 50 x 106 allogeneic bone marrow (BM)-derived MSC formulated in 4 ml infusion solution of sodium chloride supplemented with human serum albumin to be given via ultrasound-guided intra-articular injection

SUMMARY:
This open-label, single-arm, phase I/II study in mild-to-moderate stage knee osteoarthritis patients is designed to assess the safety and tolerability of intraarticular human allogeneic bone marrow-derived mesenchymal stromal cell product StromaForte. 12 male and/or female patients aged over 18 years will be enrolled. The main questions it aims to answer are:

To assess the safety and tolerability of StromaForte within 24 hours, 4 days ,28 days, 84, and 168 post injection during site visits and post injection by telephone calls. Safety and tolerability will be assessed by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs).

Eligible patients will receive one dose (50 x 106 allogeneic bone marrow (BM)-derived MSC formulated in 4 ml infusion solution (sodium chloride supplemented with human serum albumin) to be given via ultrasoundguided intra-articular injection of human allogeneic bone marrow-derived mesenchymal stromal cell product StromaForte

DETAILED DESCRIPTION:
Osteoarthritis (OA) is a severe, chronic, and progressive disease that eventually leads to disability. OA is characterized by joint pain, stiffness, limited mobility with effusion, and inflammation. It has a negative physical and psychological impact which results in a reduced quality of life. OA occurs as an imbalance between the formation and degeneration of chondrocytes and extracellular matrix which leads to progressive destruction of articular cartilage. OA symptoms were routinely managed using pharmacologic treatments including hyaluronic acid (HA) and platelet rich plasma (PRP) injections. Recent guidelines have recommended against the use of these agents. Both treatments are mainly given for pain relief and have minimal effects on stopping the progression of OA; hyaluronic acid (HA) leads to a small reduction in knee osteoarthritis pain compared with placebo, while PRP, did not result in a significant difference in symptoms or joint structure. These findings do not support broad use of them for the treatment of knee osteoarthritis.

Mesenchymal Stromal Cells (MSCs) are one of the emerging, regenerative therapies that aim to treat, prevent and even reverse OA through their immunomodulatory properties that reduce inflammation and promote angiogenesis. MSCs are proven to regulate the body's immune response in many diseases and exert anti-inflammatory effects. These immunomodulatory properties are mediated via paracrine mechanisms. Following their discovery over 50 years ago, mesenchymal stromal cells (MSCs) have become one of the most studied cellular therapeutic products by both academia and industry due to their regenerative potential and immunomodulatory properties. The promise of MSCs as a therapeutic modality has been demonstrated in a number of preclinical data as well as in clinical setting. Stromaforte cells which will be used in this study is developed within CELLCOLABS AB and were generated following the same protocol established over the last 20 years by scientists CELLCOLABS AB at the Karolinska Institute in Sweden. MSCs showed a very promising effect in patients including vocal folds, GVHD, ARDS, multiple sclerosis and recently in patients severely infected with COVID virus.

The currently completed preclinical studies on animal models showed that intra-articular injection of MSCs can promote cartilage regeneration and reduce joint inflammation to improve the OA function of joints, and no malignant transformation of MSCs has been found as well as randomized double blinded phase I/II clinical studies reported that, the clinical manifestations, radiological and histological scores of OA patients were improved, no graft-related death, tumorigenesis and infection occurred, and no serious adverse reactions were observed. These studies demonstrated safety and tolerability of the MSCs. Based on the above results preclinical and clinical studies, it is planned to conduct this study which has been designed to evaluate the safety and tolerability of intra-articular human allogeneic bone marrow-derived mesenchymal stromal cell product StromaForte in mild-to-moderate stage knee osteoarthritis patients before further clinical development.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent and comply with all procedures required by the protocol
2. Aged > 18 years at the time of signing the informed consent form
3. Diagnosed with knee OA according to American College and Rheumatology criteria and showing a stage of a mild to moderate arthritis.
4. Kellgren-Lawrence radiological classification scale II and III at screening
5. Visual analogue scale (VAS) joint pain ≥ 2.5 at screening
6. Have tried but failed conservative management including physical therapy, bracing and medications for a minimum of three months.
7. No history of prior intra-articular cortisone, hyaluronic acid, or platelet-rich plasma injection within the previous six months
8. No history of prior arthroscopic knee surgery or open knee surgery on the ipsilateral side within the past year
9. Adequate liver and renal functions with non-malignant blood profile.
10. Body Mass Index between 20 and 30 kg/m2
11. Negative for (HIV, HTLV1&2, Hep A, B, C, syphilis) infection as determined by approved serological testing
12. Negative for pregnancy as determined by a serum pregnancy test. Females of childbearing potential will be required to practice abstinence or use an effective form of contraception for 12 months following their MSC injection.
13. Fluid > 1 cm within the lateral recess of the suprapatellar pouch at the level of the superior pole of the patella with the knee extended.

Exclusion Criteria:

1. Unwilling or unable to perform any of the assessments required by the protocol
2. Patients with clinically unstable knee due to the presence of a complete anterior cruciate ligament, posterior cruciate ligament, medial collateral ligament and/or posterolateral corner tear
3. Patients with varus or valgus malalignment >5 degrees as measured by 4-foot standing antero-posterior radiographs
4. Patients with a history of a previous subtotal medial or lateral meniscectomy
5. Patients with a history of septic arthritis in the affected joint
6. Patients with a history of a prior intra-articular knee fracture
7. Severe bleeding diathesis
8. Active infection
9. Patients with unforeseen conditions that are deemed unsafe or inappropriate for the study (e.g., patients who are claustrophobic and cannot undergo an MRI) as per the discretion of the principal investigator
10. Patients with neoplasia
11. Patients participating in another clinical trial or treatment with a different investigational product within 30 days prior to inclusion in this study
12. Patients with a known history of inflammatory or rheumatic diseases such as rheumatoid arthritis

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2023-11-08 (Actual); Primary Completion 2024-11-08 (Estimated); Study Completion 2025-04-07 (Estimated)

PRIMARY OUTCOMES:
To assess safety and tolerability within 24 hours,4 days , 28, 84 and 168 days of MSC injection | From baseline to 6 months
  To assess the safety and tolerability of StromaForte within 24 hours, 4 days ,28 days, 84, and 168 post injection during site visits and post injection by telephone calls. Safety and tolerability will be assessed by reporting the number of adverse events assessed by Common Terminology Criteria For Adverse Events (CTCAE) which is the Incidence of any treatment-emergent serious adverse events (TE-SAEs), defined as the composite of death, non-fatal pulmonary embolism, stroke, hospitalization for worsening dyspnea and clinically significant laboratory test abnormalities determined per the Investigator's judgment

SECONDARY OUTCOMES:
Change from baseline in subjective pain assessment according to the VAS questionnaire 84, 168 days after treatment | From baseline to 6 months
  Change from baseline in subjective pain assessment according to the VAS questionnaire 84, 168 days after treatment. The highest pain being a number 10 on the scale and 0 the lowest.
Change from baseline in knee-joint specific function assessed by the Knee Injury and osteoarthritis outcome score (KOOS) at 84- and 168-days post-injection | From baseline to 6 months
  Change from baseline in knee-joint specific function assessed by the Knee Injury and osteoarthritis outcome score (KOOS) at 84- and 168-days post-injection. The KOOS holds five separately scored subscales: Pain, other Symptoms, Function in daily living (ADL), Function in Sport and Recreation (Sport/Rec), and knee-related Quality of Life (QOL) totalling 42 items. Pain (nine items); Symptoms (seven items); ADL Function (17 items); Sport and Recreation Function (five items); Quality of Life (four items). A Likert scale is used and all items have five possible answer options scored from 0 (No Problems) to 4 (Extreme Problems) and each of the five scores is calculated as the sum of the items included. Scores are transformed to a 0-100 scale, with zero representing extreme knee problems and 100 representing no knee problems as common in orthopaedic assessment scales and generic measures. Scores between 0 and 100 represent the percentage of total possible score achieved.
Change from baseline in arthritis pain scores using the Lequesne index assessment at 84- and 168-days post treatment | From baseline to 6 months
  Change from baseline in arthritis pain scores using the Lequesne index assessment at 84- and 168-days post treatment.
Change in Health-related quality of life according to Short-Form 12 at 168 days post-injection | From baseline to 6 months
  Change in Health-related quality of life according to Short-Form 12 at 168 days post-injection. Scores range from 0 to 100, with higher scores indicating better physical and mental health functioning.
Change in TNF-alpha in synovial fluid | From baseline to 6 months
  Change in TNF-alpha in synovial fluid from baseline to 168 days post-injection
Change in C Reactive Protein (CRP) in synovial fluid | From baseline to 6 months
  Change in C Reactive Protein (CRP) in synovial fluid from baseline to 168 days post-injection
Change in Interleukin-6 (IL-6) in synovial fluid | From baseline to 6 months
  Change in Interleukin-6 (IL-6) in synovial fluid from baseline to 168 days post-injection
Change from baseline at levels of catabolic/anabolic products of collagens | From baseline to 6 months
  Change from baseline at levels of catabolic/anabolic products of collagens in urine and/or serum at 84- and 168-days post-injection
Change from baseline level in joint space changes within the knee | From baseline to 6 months
  Change from baseline level in joint space changes within the knee using MRI at 168 days post-injection.
Change from baseline of Oxford Knee Score (OKS) | From baseline to 6 months
  Change from baseline of pain, activity, range of motion, distance…etc at 84- and 168-days post-injection using Oxford Knee Score (OKS). Score each question (item) from 0 to 4 with 0 being the worst outcome and 4 being the best outcome. The scores are then summed to produce an overall score running from 0 (worst possible) to 48 (best outcome).

OTHER OUTCOMES:
Change from baseline of cell composition of blood and synovial fluids | From baseline to 6 months
  Change from baseline of cell composition of blood and synovial fluids at 168-days post-injection

CONTACTS AND LOCATIONS:
Overall Officials: Fahti Yousef, PhD, Principal Investigator — Cellcolabs Clinical SPV Limited
Locations (1):
- Burjeel Medical City, Abu Dhabi, United Arab Emirates

IPD SHARING:
Plan to Share IPD: Undecided